CLINICAL TRIAL: NCT03927482
Title: C.A.R.E.S.: A Mobile Health Program for Alcohol Risk Reduction for an Under- Served College Population
Brief Title: CARES: A Mobile Health Program for Alcohol Risk Reduction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Beth Bock, Ph.D., Senior Research Scientist, The Miriam Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 7147117; R42AA026788 (NIH)
Record Dates: First submitted 2019-04-23; First posted 2019-04-25 (Actual); Results first posted 2022-08-31 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Alcohol Abuse
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Assessors will be blind to the participant's randomization assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CARES mobile app (Experimental): Participants in this arm will receive 12 weeks of text messages and use of the smart phone mobile app that provides support for alcohol risk reduction.
  Interventions: Behavioral: CARES mobile smart phone app
- Alcohol Education (Active Comparator): Those randomized to the control arm will be given access to an online alcohol education intervention; Check Your Drinking (CYD: www.CheckYourDrinking.net). CYD provides normative feedback on the user's drinking habits relative to his/her peers.
  Interventions: Behavioral: Check Your Drinking

INTERVENTIONS:
Behavioral: CARES mobile smart phone app — The CARES smart phone mobile app contains a number of features to support safety while drinking and reduced alcohol consumption plus regular test messages for personal support
  Arms: CARES mobile app
Behavioral: Check Your Drinking — Check Your Drinking is an online alcohol assessment that provides normative feedback on the user's drinking habits relative to his/her peers. Alcohol interventions that provide normative feedback are rated by the NIAAA Alcohol Intervention Matrix as effective and low cost, and with few administrative or structural barriers to implementation thus making it suitable for community colleges.
  Arms: Alcohol Education

SUMMARY:
In this fast-track STTR, Phase 1 will develop and test a mobile phone app among 40 adult community college students. The app is designed to reduce risky drinking behaviors and improve user safety. In Phase 2 the app ("CARES") will be tested with 200 adult community college students who drink alcohol. Participants will be randomly assigned to the "CARES" app or an alcohol education control condition and will use the app for 12 weeks. Six month outcomes will assess changes in drinking related behaviors.

DETAILED DESCRIPTION:
This STTR builds on our successful pilot that developed a text message-delivered alcohol intervention for, and in collaboration with CCS. Phase I will develop and test a smart phone application (the "Cares" app) incorporating the text message program with additional features and functionality requested by students in the pilot trial (Aim 1.1). After obtaining user feedback (Aim 1.2) programming will be completed in both iOS and Android languages. To ensure that the College Alcohol Risk Education System (CARES) is well positioned to get into the community college marketplace, it is critical to demonstrate efficacy. Phase 2 will conduct an efficacy trial of CARES compared to a competing alcohol education program that would be feasible for most community colleges to adopt, thus providing a real-world comparison with data suitable to support future efforts toward commercialization. This study will also identify the types of individuals for whom CARES is more/less effective and identify how it might be improved.

ELIGIBILITY:
Inclusion Criteria:

* Currently enrolled community college student
* At least 2 heavy drinking episodes in past 2 weeks at recruitment
* Own smart phone

Exclusion Criteria:

* Alcohol abuse disorder or currently in treatment for alcohol-related problems

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 239 (Actual)
Dates: Start 2018-08-02 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2022-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beth C Bock, PhD, Principal Investigator — The Miriam Hospital
Locations (1):
- The Miriam Hospital- CORO building, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bock B, Deutsch C, Dunsiger S, Rosen RK, Walaska K, Lantini R, Foster R. C.A.R.E.S: A mobile health program for alcohol risk reduction in community college students. Contemp Clin Trials. 2021 Aug;107:106493. doi: 10.1016/j.cct.2021.106493. Epub 2021 Jun 26. PMID 34182157

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CARES Mobile App | Alcohol Education
Started | 118 | 121
Completed | 110 | 115
Not Completed | 8 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CARES Mobile App | Alcohol Education | Total
Number analyzed (Participants) | 118 | 121 | 239
Age, Continuous [Mean (Standard Deviation); unit: Years] | 22.9 (3.2) | 22.9 (3.3) | 22.9 (3.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 85 | 168
  Male | 35 | 36 | 71
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23 | 21 | 44
  Not Hispanic or Latino | 95 | 100 | 195
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 12 | 8 | 20
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 25 | 25 | 50
  White | 63 | 80 | 143
  More than one race | 11 | 5 | 16
  Unknown or Not Reported | 6 | 3 | 9
Region of Enrollment [Number; unit: participants]
  United States | 118 | 121 | 239
Drinks per week [Mean (Standard Deviation); unit: drinks] | 7.81 (7.24) | 7.78 (6.62) | 7.79 (6.93)
Binge Drinking Days [Mean (Full Range); unit: days] | 0.86 [0 to 7] | 0.88 [0 to 4] | 0.87 [0 to 7]

OUTCOME MEASURES:

1. Primary Outcome: Drinks Per Week
Description: Average drinks based on 30 day timeline follow back of all alcohol consumption
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: drinks
Arm/Group | CARES Mobile App | Alcohol Education
Number analyzed (Participants) | 118 | 121
drinks | 4.05 (4.83) | 5.58 (6.29)

2. Primary Outcome: Alcohol Related Consequences
Description: Negative life events related to drinking assessed by the Brief Young Adult Alcohol Consequences Questionnaire. Calculates a total score from 0-48, with higher numbers indicating worse outcomes.
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CARES Mobile App | Alcohol Education
Number analyzed (Participants) | 118 | 121
score on a scale | 4.34 (5.94) | 4.95 (6.12)

3. Secondary Outcome: Situational Confidence
Description: Confidence in drinking resistance assessed by the Brief Situational Confidence Questionnaire. Scores 8 items from 0% to 100% confidence with higher scores indicating better confidence.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CARES Mobile App | Alcohol Education
Number analyzed (Participants) | 118 | 121
score on a scale | 72.6 (21.4) | 74.6 (19.6)

4. Secondary Outcome: Protective Strategies
Description: Skills in using alcohol-protective behaviors measured by the Protective Behavioral Strategies Survey. A 15-item survey, each item is scored from 0 to 6 to indicate use of behavioral strategies and the total score is a sum of all items. Higher scores indicate more (better) use of protective strategies.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CARES Mobile App | Alcohol Education
Number analyzed (Participants) | 118 | 121
score on a scale | 3.65 (0.69) | 3.48 (0.73)

ADVERSE EVENTS:
Time Frame: 1 year
Description: This is a low-risk behavioral intervention providing educational information on risks of alcohol consumption.
Arm/Group | CARES Mobile App | Alcohol Education
All-Cause Mortality (participants affected / at risk) | 0/118 | 0/121
Serious Adverse Events (participants affected / at risk) | 0/118 | 0/121
Other Adverse Events (participants affected / at risk) | 0/118 | 0/121

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-12-17): https://cdn.clinicaltrials.gov/large-docs/82/NCT03927482/Prot_SAP_000.pdf
  • Informed Consent Form (2020-12-28): https://cdn.clinicaltrials.gov/large-docs/82/NCT03927482/ICF_001.pdf